CLINICAL TRIAL: NCT03728621
Title: Individual Versus Group-based Lifestyle Intervention in Obese Children: Effects on Anthropometry and Metabolic Profile
Brief Title: Lifestyle Interventions and Metabolic Profile in Obese Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Elvira Verduci, MD PhD Assistant professor in Pediatrics, University of Milan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 139/2010/CE
Record Dates: First submitted 2018-10-22; First posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Childhood Obesity; Obesity; Pediatric Obesity; Dyslipidemias; Cardiovascular Risk Factor; Life Style
Keywords: obesity; child; AIP; lifestyle intervention
MeSH Terms: conditions — Pediatric Obesity; Obesity; Dyslipidemias | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This is a randomized, prospective, controlled study of 12 months a total of 170 children were consecutively recruited among those with diagnosis of obesity (in accordance with World Health Organization (WHO) criteria) by primary care pediatricians and admitted to the Department of Pediatrics, San Paolo Hospital, Milan, Italy, between January 2012 and June 2017. Inclusion criteria were: age at recruitment ≥6 years; weight at birth ≥2500 g and <4000 g; gestational age 37-42 weeks; single birth; Caucasian race; family residing in Milan or neighborhood (≤30 km). Children having syndromic, organic and hormonal conditions besides obesity were excluded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual-based lifestyle intervention (Experimental): Promotion of normocaloric & balanced diet and physical activity
  Interventions: Behavioral: Normocaloric and balanced diet, physical activity
- Group-based lifestyle intervention (Experimental): Promotion of normocaloric & balanced diet and physical activity
  Interventions: Behavioral: Normocaloric and balanced diet, physical activity

INTERVENTIONS:
Behavioral: Normocaloric and balanced diet, physical activity — Promotion of normocaloric & balanced diet and physical activity

SUMMARY:
This study evaluates if promotion of a normocaloric and balanced diet and of physical activity, through an individual- or group-based lifestyle intervention of 12 months, may affect anthropometric measurements and metabolic profile in obese children.

DETAILED DESCRIPTION:
Obese children are at risk of metabolic and cardiovascular complications both during pediatric age and later and they often show components of metabolic syndrome, such as dyslipidemia, hypertension and disturbed glucose metabolism . These complications are strictly associated with insulin resistance/hyperinsulinemia which is one of the most important contributing factors to cardiovascular disease. The gold standard technique to determine whole-body insulin sensitivity, the hyperinsulinemic-euglycemic clamp, is expensive, invasive and requires considerable expertise to be performed. Therefore, several surrogate measures have been developed. Among these, the triglyceride-glucose index (TyG) is a useful indicator, providing an easily and widely available simple laboratory method as a surrogate to estimate insulin resistance in adult, children and adolescents. Other useful indicators of insulin resistance and insulin sensitivity are the homeostatic model assessment of insulin resistance (HOMA-IR) and the quantitative insulin sensitivity check (QUICK) index, respectively, while HOMA-β% is useful to evaluate pancreatic β-cell function.

Among cardiovascular complications, obesity-related atherogenic dyslipidemia is a risk factor for cardiovascular disease. In childhood, atherogenic dyslipidemia may be associated with structural and functional vascular changes, as increased carotid intima-media thickness and increased arterial stiffness. The atherogenic index of plasma (AIP) is a recognized valuable indicator of the size of pre- and anti-atherogenic lipoprotein particle and is considered a major predictive marker of atherosclerosis risk. Additionally, it might be more promising than other lipid variables in assessing cardiovascular risk.

Guidelines for treatment of childhood obesity recommend intensive lifestyle interventions, involving diet, physical activity and behavior change, in an age-appropriate manner. While it is recognized that these interventions could favorably influence some variables of metabolic profile of obese children, no study has reported accurate possible effect on triglyceride-glucose index and atherogenic index of plasma. Furthermore, pediatric obesity interventions may be group and/or individual-based. The group-based intervention requires less resources, children may benefit from a positive social environment, but the attention to individual needs is limited, which may weaken outcomes. On the other hand, the individual-based intervention allows to tailor dietary and physical counselling on individual's needs but is more expensive and requires greater resources.

The aims of the study are to establish in patients who undergone individual versus group based intervention:

1. Effect on adiposity measured by BMI-zScore
2. effect on gluco-insulin metabolism evaluated by homa-index
3. effect on lipid profile evaluated by aterogenic index (AIP)

ELIGIBILITY:
Inclusion Criteria:

* Obesity confirmed by BMI z-score >2 according to WHO growth charts
* Age at recruitment ≥6 years
* weight at birth ≥2500 g and <4000 g
* gestational age 37-42 weeks
* single birth
* Caucasian ethny
* family residing in Milan or neighborhood (≤30 km)

Exclusion Criteria:

* Syndromic, organic and hormonal conditions besides obesity
* Age at recruitment <6 years
* Low birthweight (<2500 g), birthweight >4000 g
* Pre-term or post-term birth
* Twin delivery
* Other ethnies than Caucasian

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Height | 0 (t0)-12 months (t1)
  Expressed in meters
Blood levels of total cholesterol | 0 (t0)-12 months (t1)
Weight | 0 (t0)-12 months (t1)
  Expressed in Kilograms
Body Mass Index (BMI) | 0 (t0)-12 months (t1)
  Expressed in kg/m^2
Waist-to-height ratio | 0 (t0)-12 months (t1)
  The ratio between waist circumference (cm) and height (cm)
Waist circumference | 0 (t0)-12 months (t1)
  Expressed in cm
Triceps Skinfold Thickness | 0 (t0)-12 months (t1)
  Expressed in mm, measured with an accurate plicometer
Tanner Stage | 0 (t0)-12 months (t1)
  Classification of sexual maturation according to Tanner criteria
Blood levels of LDL cholesterol | 0 (t0)-12 months (t1)
Blood levels of HDL cholesterol | 0 (t0)-12 months (t1)
Blood levels of triglycerides | 0 (t0)-12 months (t1)
Blood levels of apolipoprotein A1 (ApoA1) | 0 (t0)-12 months (t1)
Blood levels of apolipoprotein B (ApoB) | 0 (t0)-12 months (t1)
Blood levels of insulin | 0 (t0)-12 months (t1)
Blood levels of glucose | 0 (t0)-12 months (t1)
HOmeostatic Model Assessment of Insulin Resistance (HOMA-IR) | 0 (t0)-12 months (t1)
  calculated as the product of fasting glucose (mmol/L) and fasting insulin (U/mL) divided by 22.5
QUantitative Insulin sensitivity ChecK (QUICK) index | 0 (t0)-12 months (t1)
  1/[log10 fasting plasma insulin (U/mL) + log10 glucose (mg/dL)]
HOMA-β% | 0 (t0)-12 months (t1)
  [20 fasting insulin in (U/mL)/(fasting glucose (mmol/L) - 3.5]
Triglyceride-Glucose index (TyG index) | 0 (t0)-12 months (t1)
  ln[fasting triglycerides (mg/dL) fasting glucose (mg/dL)/2]
Atherogenic Index of Plasma (AIP) | 0 (t0)-12 months (t1)
  log10 of the ratio of plasma triglycerides to HDL-cholesterol

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Paolo, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Verduci E, Banderali G, Di Profio E, Vizzuso S, Zuccotti G, Radaelli G. Effect of individual- versus collective-based nutritional-lifestyle intervention on the atherogenic index of plasma in children with obesity: a randomized trial. Nutr Metab (Lond). 2021 Jan 13;18(1):11. doi: 10.1186/s12986-020-00537-w. PMID 33436021